CLINICAL TRIAL: NCT04492787
Title: A Randomized,double-blind,placebo-controlled,multicenter Study to Evaluate the Efficacy and Safety of Changkang Granule in the Treatment of Diarrhea-predominant Irritable Bowel Syndrome (IBS-D)
Brief Title: Efficacy and Safety of Changkang Granule in the Treatment of Diarrhea-predominant Irritable Bowel Syndrome (IBS-D)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-TCM-CKKL-Ⅱ
Record Dates: First submitted 2020-07-23; First posted 2020-07-30 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Irritable Bowel Syndrome with Diarrhea
Keywords: Changkang Granule

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Changkang Granules (Experimental): Changkang Granules
  Interventions: Drug: Changkang Granule
- Changkang Placebo Granules (Placebo Comparator): Changkang Placebo Granules
  Interventions: Drug: Changkang Placebo Granule

INTERVENTIONS:
Drug: Changkang Granule — Take Changkang granule before meals twice a day , one bag for each time
  Arms: Changkang Granules
Drug: Changkang Placebo Granule — Take Changkang Placebo granule before meals twice a day , one bag for each time
  Arms: Changkang Placebo Granules

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of Changkang granule as compared to placebo over a 8-week treatment period and explore TCM syndrome types.

DETAILED DESCRIPTION:
The clinical phase of the study comprises up to 2 weeks of screening for patient's eligibility, a 2-week run-in period , a 8-week double-blind treatment period, and a 4-week safety follow-up.

Patients report their IBS-related symptoms daily from run-in until end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The patients with diarrhea predominant irritable bowel syndrome (IBS-D) met Rome IV criteria;
2. It is in accordance with the syndrome differentiation standard of TCM, such as the syndrome of liver Qi multiplying spleen, spleen stomach weakness, spleen kidney yang deficiency or large intestine damp heat syndrome;
3. Male or female aged 18 to 65 years (including the boundary value);
4. The weekly mean NRS score of abdominal pain was ≥ 3.0, and the number of days with stool type 6 or 7 was more than 2 days per week;
5. IBS-SSS score>175;
6. Signed informed consent voluntarily.

Exclusion Criteria:

1. Patients with IBS-C、IBS-M or IBS-U；
2. Those who had been diagnosed with organic diseases of digestive system, such as inflammatory bowel disease, intestinal tuberculosis, intestinal tumor, etc., or still combined with peptic ulcer and infectious diarrhea;
3. Patients were diagnosed with similar symptoms of irritable bowel syndrome in the past, such as eosinophilic enteritis, collagen enteritis, lactose intolerance, etc;
4. Patients with non intestinal diseases of digestive system, such as tuberculous peritonitis, gallstones, liver cirrhosis, chronic pancreatitis, etc;
5. Previous diagnosis of systemic diseases affecting gastrointestinal function, such as hyperthyroidism or hypothyroidism, endometriosis, chronic renal insufficiency, autoimmune diseases, diabetes, etc
6. With history of abdominal surgery (e.g., cholecystectomy);
7. Patients with severe cardiovascular disease, liver, kidney and other major organ diseases, hematopoietic system diseases, tumor, nervous or mental system diseases (such as severe depression, severe anxiety)
8. Those who could not stop using concomitant drugs (prokinetic agents, anticholinergics, calcium channel blockers, 5-HT3 receptor antagonists, antidiarrheal agents, antacids, antidepressants, antianxiety drugs, intestinal flora regulators, etc.) that affected gastrointestinal motility and function ;
9. Taking emergency medication in the run-in period；
10. Pregnant or lactating women；
11. Those who are allergic to the test drug, emergency drug and its ingredients；
12. Suspected or confirmed history of alcohol and drug abuse;
13. Patients who participated in other clinical trials within one month before enrollment;
14. The researchers believe that others are not suitable for clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Are Composite Responders Consistency Scores | 8 week
  Composite responders are defined as participants who met the weekly response criteria for at least 50% of the weeks with diary entries over the 8-week interval.
  The patient will be considered a weekly responder if she/he meets both of the following criteria in the same week.
  1. Abdominal pain response: decrease in weekly average of worst abdominal pain score in the past 24 hours of at least 30% compared with baseline;
  2. Stool consistency response: decrease of at least 50% in the number of days per week with at least one stool that has a consistency of Type 6 or 7 compared with baseline.

SECONDARY OUTCOMES:
Percentage of Participants Who Are Responders in Abdominal Pain Scores | 8 week
  Abdominal pain responders are defined as participants who met the weekly response criteria for at least 50% of the weeks with diary entries over the 8-week interval; Weekly response: decrease in weekly average of worst abdominal pain score in the past 24 hours of at least 30% compared with baseline.
Percentage of Participants Who Are Responders in Stool Consistency Scores | 8 week
  Stool consistency responders are defined as participants who met the weekly response criteria for at least 50% of the weeks with diary entries over the 8-week interval.
  Weekly response: decrease of at least 50% in the number of days per week with at least one stool that has a consistency of Type 6 or 7 compared with baseline.
Change from baseline to each week during follow up for IBS-symptoms abdominal pain； | 8 week
  Abdominal Pain：Scored between 0 and 10 (none to severe).
Change from baseline to each week during follow up for IBS-symptoms stool consistency; | 8 week
  Stool consistency：Bristol Stool Scale（Scored 1-7）.
Change from baseline to each week during follow up for IBS-symptoms bloating | 8 week
  Bloating：Scored between 0 and 10.
Change from baseline to each week during follow up for IBS-symptoms urgency | 8 week
  The change of frequency of defecation urgency per week compared with baseline.
Change from baseline to each week during follow up for IBS-symptoms Defecation frequency | 8 week
  Change from baseline in mean number of bowel movements per week.
Disappearance rate of traditional Chinese Medicine（TCM）symptom | 8 week
  Each syndrome type has 2-3 symptoms，liver Qi multiplying spleen syndrome includes Chest and flank fullness, depression, irritability

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Xiyuan Hospital, China Academy of Traditional Chinese Medicine, Beijing
  - Shengjing Hospital of China Medical University, Dalian
  - Gansu Provincial Hospital of TCM, Gansu
  - The first affiliated Hospital of Hunan University of Traditional Chinese Medicine, Hunan
  - Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai
  - West China Hospital of Sichuan University, Sichuan
  - Wenzhou Hospital of Traditional Chinese Medicine, Wenzhou
  - Xiamen Hospital of Traditional Chinese Medicine, Xiamen

IPD SHARING:
Plan to Share IPD: No